CLINICAL TRIAL: NCT06788717
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Comprehensive® Primary Revision Stems (Implants and Instrumentation) - A Retrospective and Prospective Consecutive Series Study
Brief Title: MDR - Comprehensive Primary Revision Stems PMCF
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-50E
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Pain; Shoulder Injuries; Shoulder Fractures; Shoulder Disease; Shoulder Arthritis
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Shoulder Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: The study population will comprise a consecutive cohort of 59 cases (males and females), implanted with the Comprehensive Primary Revision Stem.
  Interventions: Device: Comprehensive Primary Revision Stems

INTERVENTIONS:
Device: Comprehensive Primary Revision Stems — Comprehensive Primary Revision Stem (implants and instrumentation) when used for shoulder arthroplasty.

SUMMARY:
The objective of this retrospective and prospective consecutive series PMCF (Post Market Clinical Follow Up) study is to collect long-term data confirming safety, performance and clinical benefits of the Comprehensive Primary Revision Stems (implants and instrumentation) when used for shoulder arthroplasty at 1, 3, 5, 7 and 10 years.

DETAILED DESCRIPTION:
The safety of this device will be assessed by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The performance will be evaluated by assessment of reported clinical outcome measures (PROMs) as well as radiographic outcomes.

ELIGIBILITY:
Inclusion Criteria

* Patient must be 18 years of age or older.
* Patient must be willing and able to follow directions.
* Study devices must have been implanted following the surgical technique and IFU for the Comprehensive Revision Stem

Exclusion Criteria

* Off-label use.
* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent.
* Patient is unwilling to sign informed consent.
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of subjects implanted with the Comprehensive Primary Revision Stems according to the approved indications will be identified and invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship at 10 years follow-up (Kaplan Meier) | 10 years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method.
Frequency and Incidence of Adverse Events (Safety) | 10 years
  Monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Western Ontario Arthritis of the Shoulder (WOOS) outcome measure. | 10 years
  The secondary objective is the assessment of performance and clinical benefits by recording patient reported clinical outcome measures (PROMs), through the use of the Western Ontario Osteoarthritis of the Should Score (WOOS). The WOOS is a 19 item questionnaire. Patients rate their symptoms from no pain extreme pain. The total score is calculated where 0 is a normal healthy shoulder and 1900 is the worst possible result. WOOS% (% of raw score) can be calculated using the formula (1900 - the score)/19 and then 0% is the worst possible result and 100% is the best possible result.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, MBA, Study Director — Zimmer Biomet
Locations (2):
- Cedars Sinai Medical Center, Los Angeles, California, United States
- Aalborg University Hospital, Aalborg, Denmark